CLINICAL TRIAL: NCT01500473
Title: Therapeutic Effect of Desogestrel on Ventilatory Control in Patients With Congenital Central Hypoventilation Syndrome
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Only one subject was studied, who did not respond.
Sponsor: Children's Hospital Los Angeles (Other)
Responsible Party: Principal Investigator, Iris Perez, Principal Investigator, Children's Hospital Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCI-11-00057
Record Dates: First submitted 2011-12-22; First posted 2011-12-28 (Estimated); Results first posted 2023-09-28 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-10

CONDITIONS: Congenital Central Hypoventilation Syndrome
MeSH Terms: conditions — Congenital central hypoventilation syndrome | interventions — Desogestrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Females with CCHS > 16 years old on desogestrel (Experimental): open label studied on drug.
  Interventions: Drug: Desogestrel

INTERVENTIONS:
Drug: Desogestrel — Reclipsen oral contraceptive pill with 0.03mg ethinyl estradiol and 0.15mg desogestrel
  Other Names: Reclipsen

SUMMARY:
Background: Congenital Central Hypoventilation Syndrome (CCHS) is a rare disorder of automatic control of breathing. This disease can manifest as early as birth. Patients with this disease have a fundamental lack of central drive breathing. They do not mount any responses to hypoxia or hypercapnia during sleep or wakefulness. This places them at risk of injury or death whenever they are not consciously breathing. They require lifelong assisted ventilation while sleeping, and some while awake. Progesterone is a known respiratory stimulant in normal individuals, and it has been shown in one study of 2 patients that this drug may improve CO2 responsiveness in patients with CCHS. However, this observation requires confirmation.

Hypothesis: Exogenous progesterone (in oral contraception pills) will improve CO2 responsivity by hyperoxic hypercapnic ventilatory response testing, hypoxic responsivity using 5-breath nitrogen breathing, hyperoxic ventilatory response while breathing 100% oxygen, and improve spontaneous ventilation during sleep in CCHS females >15-years of age. The progesterone will also depress ventilatory response using a hyperoxia test.

Study Methodology: Baseline measures of CO2 and oxygen responsivity, and spontaneous ventilation during sleep, will be performed at baseline and after 3-weeks of taking a progesterone containing oral contraceptive agent. CO2 responsivity will be measured using a hyperoxic hypercapnic ventilatory response test. Hypoxic responsivity will be measured using a 5-breath 100% nitrogen breathing test. Hyperoxic responsivity will be measured by having subjects breathe 100% oxygen for 2-minutes. Subjects will perform an overnight polysomnogram to assess adequacy of gas exchange during spontaneous breathing while asleep. A progesterone containing oral contraception pill will then be given for 3-weeks, and the above measures repeated. Serum progesterone will be measured at baseline and at the time of study.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed congenital central hypoventilation syndrome (CCHS)
* female
* greater than or equal to 16 years of age

Exclusion Criteria:

* less than 16 years of age
* male
* pregnant
* poor adherence to medications
* inability to perform pulmonary maneuvers for tests
* contraindications to oral contraceptives
* pulmonary hypertension

Ages: 16 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1 (Actual)
Dates: Start 2012-02 (Actual); Primary Completion 2016-05-11 (Actual); Study Completion 2016-05-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Iris Perez, MD, Principal Investigator — Children's Hospital Los Angeles
Locations (1):
- Children's Hospital Los Angeles, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Females With CCHS > 16 Years Old on Desogetrel: open label studied on drug.
  Desogestrel: Reclipsen oral contraceptive pill with 0.03mg ethinyl estradiol and 0.15mg desogestrel
Period: Overall Study
Arm/Group | Females With CCHS > 16 Years Old on Desogetrel
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Females With CCHS > 16 Years Old on Desogetrel
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Hypoxic Ventilatory Response
Description: Increase in minute ventilation as oxygen saturation of hemoglobin falls.
Time Frame: 3 weeks
Measure: Number; unit: subjects with positive response
Arm/Group | Females With CCHS > 16 Years Old on Desogetrel
Number analyzed (Participants) | 1
subjects with positive response | 0

2. Primary Outcome: Hypercapnic Ventilatory Response
Description: Increase in ventilation with increasing partial pressure of CO2
Time Frame: 3 weeks
Measure: Number; unit: liters per minute/ mmHg PCO2
Arm/Group | Females With CCHS > 16 Years Old on Desogestrel
Number analyzed (Participants) | 1
liters per minute/ mmHg PCO2 | -0.520

3. Primary Outcome: Time Maintained Ventilation Off Mechanical Ventilation During Sleep.
Description: length of time the subject could breathe adequately spontaneously until SpO2 fell below 80% and or PetCO2 rose above 65 mmHg.
Time Frame: 3 weeks
Measure: Number; unit: seconds
Arm/Group | Females With CCHS > 16 Years Old on Desogestrel
Number analyzed (Participants) | 1
seconds | 89

ADVERSE EVENTS:
Arm/Group | Females With CCHS > 16 Years Old on Desogetrel
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed. Only one subject was enrolled.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes